CLINICAL TRIAL: NCT04541888
Title: A Phase 3, Multicenter, Randomized, Double-blind, Vehicle-controlled Efficacy and Safety Study of CsA Ophthalmic Gel in Subjects With Moderate to Severe Dry Eye Disease
Brief Title: Assess the Safety and Efficacy of CsA Ophthalmic Gel in Subjects With Moderate to Severe Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKY-CSA-202001
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): 322 subjects will be treated with CsA eye gel: 0.3 g: 0.15 mg, 1 times daily, The treatment period is 12 weeks. The basic medicine is Hypromellose Eye Drops, 3 times daily for 12 weeks.
  Interventions: Drug: CsA Ophthalmic Gel; Drug: Hypromellose Eye Drop
- Control group (Placebo Comparator): 322 subjects will be treated with Placebo : 0 g: 0mg, 1 times daily, The treatment period is 12 weeks. The basic medicine is Hypromellose Eye Drops, 3 times daily for 12 weeks.
  Interventions: Drug: Placebo; Drug: Hypromellose Eye Drop

INTERVENTIONS:
Drug: CsA Ophthalmic Gel — The CsA eye gel of 0.3 g: 0.15 mg
  Other Names: CsA gel
  Arms: Experimental Group
Drug: Placebo — Placebo
  Arms: Control group
Drug: Hypromellose Eye Drop — Hypromellose Eye Drops of 10ml：50mg, 3 times daily, 1-2 drop
  Other Names: zhenshishuang

SUMMARY:
The purpose of this study is to explore the efficacy and safety of CsA ophthalmic gel in the treatment of moderate to severe dry eye disease .

DETAILED DESCRIPTION:
A multicenter,randomized, double-blind, vehicle-controlled Study.Subjects will be randomly assigned to the experimental group and the control group,experimental group: CsA eye gel: 0.3 g: 0.15 mg, once daily;One drop into each eye when you use it.hypromellose eye drops:10ml：50mg,three times a day Control group: vehicle. One drop into the eye, once daily;One drop into each eye when you use it.hypromellose eye drops:10ml：50mg,three times a day

ELIGIBILITY:
Inclusion Criteria:

1）18≤Age≤80, both male and female 2）According to the symptoms and signs and ophthalmologic examinations, the patients were diagnosed as moderate to severe dry eye

1. EDS score is more than 40 points;
2. BUT is less than 10 s;
3. Schirmer test result is less than 10mm/5 min;
4. ICSS≥2 points. 3）The ICSS score of baseline decreased by≤ 20% compared with that of screening period 4）Agree to participate in the study and voluntarily sign informed consent.

Exclusion Criteria:

1. Severe dry eye patients requiring surgical treatment
2. Had inner eye surgery within 12 months prior to screening or required inner eye surgery during the study period;Eyelid surgery was performed within 6 months prior to screening
3. Patients receiving permanent lacrimal insertion or patients receiving temporary lacrimal insertion within 6 months prior to screening;
4. Operation-induced dry eye
5. Glaucoma patients;
6. Unwilling to avoid wearing contact lenses;
7. Systemic inflammation or active eye infection and blepharitis;
8. Patients with multiple episodes of viral keratitis
9. Patients with ocular cicatricial pemphigoid, obvious conjunctival scar, ocular chemical burn and neurotrophic keratoconjunctivitis
10. Patients with malignant tumors in the past 5 years, except the thoroughly cured basal cell carcinoma of skin, squamous cell carcinoma in situ of skin, and primordial cervical cancer;
11. Perimenopausal women are taking hormone replacement therapy
12. Patients who cannot stop using other eye drops and other ophthalmic preparations during the study period;
13. Patients with severe cardiopulmonary diseases, uncontrolled hypertension and diabetes, etc. that affect the collection or compliance of study parameters;
14. ALT and AST ≥ 2 times of the normal upper limit, and serum creatinine ≥ 1.5 times of the normal upper limit
15. With a history of central nervous system disease or epilepsy, and/or a mental state that does not cooperate
16. Pregnant women and lactating women, or women of childbearing age, do not adopt effective contraceptive measures;
17. Participated in other clinical trials or participated in other clinical trials within 1 months before the election;
18. Systemic or topical cyclosporine drugs within 1 months before the election;
19. Allergy to CsA, fluorescein or any component of the drug is known；
20. Patients who were not considered suitable for the study, including those who were unable or unwilling to comply with the protocol requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Proportion of patients whose corneal fluorescein staining score (ICSS) decreased by ≥1 point from baseline at visit 5 (study eye) | 84 days after admission
  ICSS：no staining = 0，few/rare punctate lesions = 1，discrete and countable lesions = 2，lesions too numerous to count，but not coalescent = 3，coalescent = 4

SECONDARY OUTCOMES:
EDS score at the NO.3, NO.4 and NO.5 visit was compared with the baseline EDS score (binocular) | 14 days after admission ，42 days after admission ，84days days after admission
  0-100 points VAS score was evaluated
Average changes in VAS scores of 6 dry eye symptoms (burning/needling sensation, pruritus, foreign body sensation, discomfort, photophobia and pain) at the NO.3, NO.4 and NO.5 visit were compared with baseline (binocular) | 14 days after admission ，42 days after admission ，84days days after admission
  0-100 points VAS score was evaluated
corneal fluorescein staining score (ICSS)at the NO.3, NO.4 and NO.5 visit was compared with the baseline (binocular) | 14 days after admission ，42 days after admission ，84days days after admission
  ICSS：no staining = 0，few/rare punctate lesions = 1，discrete and countable lesions = 2，lesions too numerous to count，but not coalescent = 3，coalescent = 4
oxford score at the NO.3, NO.4 and NO.5 visit was compared with the baseline (binocular) | 14 days after admission ，42 days after admission ，84days days after admission
  0~V grade was evaluated
Tear break-up time(BUT) at the NO.3, NO.4 and NO.5 visit was compared with the baseline (binocular) | 14 days after admission，42 days after admission ，84days days after admission
  The time taken for the first dry spot to appear on the cornea after a complete blink with fluorescein
Schirmer's II test (with anesthetic) at the NO.3, NO.4 and NO.5 visit was compared with the baseline (binocular) | 14 days after admission ，42 days after admission ，84days days after admission
  Basal tear secretion with topical anesthesia, determined by the moisture length on the filter paper in 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: shiyou zhou, PHD, Study Director — Ophthalmological Center of Zhongshan University
Locations (1):
- Ophthalmological Center of Zhongshan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Utine CA, Stern M, Akpek EK. Clinical review: topical ophthalmic use of cyclosporin A. Ocul Immunol Inflamm. 2010 Oct;18(5):352-61. doi: 10.3109/09273948.2010.498657. PMID 20735287
- [Result] Kunert KS, Tisdale AS, Gipson IK. Goblet cell numbers and epithelial proliferation in the conjunctiva of patients with dry eye syndrome treated with cyclosporine. Arch Ophthalmol. 2002 Mar;120(3):330-7. doi: 10.1001/archopht.120.3.330. PMID 11879137
- [Result] Strong B, Farley W, Stern ME, Pflugfelder SC. Topical cyclosporine inhibits conjunctival epithelial apoptosis in experimental murine keratoconjunctivitis sicca. Cornea. 2005 Jan;24(1):80-5. doi: 10.1097/01.ico.0000133994.22392.47. PMID 15604871
- [Result] Perry HD, Doshi-Carnevale S, Donnenfeld ED, Solomon R, Biser SA, Bloom AH. Efficacy of commercially available topical cyclosporine A 0.05% in the treatment of meibomian gland dysfunction. Cornea. 2006 Feb;25(2):171-5. doi: 10.1097/01.ico.0000176611.88579.0a. PMID 16371776
- [Result] Leonardi A, Messmer EM, Labetoulle M, Amrane M, Garrigue JS, Ismail D, Sainz-de-la-Maza M, Figueiredo FC, Baudouin C. Efficacy and safety of 0.1% ciclosporin A cationic emulsion in dry eye disease: a pooled analysis of two double-masked, randomised, vehicle-controlled phase III clinical studies. Br J Ophthalmol. 2019 Jan;103(1):125-131. doi: 10.1136/bjophthalmol-2017-311801. Epub 2018 Mar 15. PMID 29545413
- [Result] Kim EC, Choi JS, Joo CK. A comparison of vitamin a and cyclosporine a 0.05% eye drops for treatment of dry eye syndrome. Am J Ophthalmol. 2009 Feb;147(2):206-213.e3. doi: 10.1016/j.ajo.2008.08.015. Epub 2008 Oct 9. PMID 18848318
- [Result] Holland EJ, Luchs J, Karpecki PM, Nichols KK, Jackson MA, Sall K, Tauber J, Roy M, Raychaudhuri A, Shojaei A. Lifitegrast for the Treatment of Dry Eye Disease: Results of a Phase III, Randomized, Double-Masked, Placebo-Controlled Trial (OPUS-3). Ophthalmology. 2017 Jan;124(1):53-60. doi: 10.1016/j.ophtha.2016.09.025. Epub 2016 Oct 27. PMID 28079022
- [Result] Tauber J, Karpecki P, Latkany R, Luchs J, Martel J, Sall K, Raychaudhuri A, Smith V, Semba CP; OPUS-2 Investigators. Lifitegrast Ophthalmic Solution 5.0% versus Placebo for Treatment of Dry Eye Disease: Results of the Randomized Phase III OPUS-2 Study. Ophthalmology. 2015 Dec;122(12):2423-31. doi: 10.1016/j.ophtha.2015.08.001. Epub 2015 Sep 11. PMID 26365210
- [Result] Bron AJ, Evans VE, Smith JA. Grading of corneal and conjunctival staining in the context of other dry eye tests. Cornea. 2003 Oct;22(7):640-50. doi: 10.1097/00003226-200310000-00008. PMID 14508260